CLINICAL TRIAL: NCT06219759
Title: Reinnervation and Neuromuscular Transmission in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Reinnervation and Neuromuscular Transmission in ALS
Acronym: RANTAL
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 8340; 1-10-72-153-23 (Other: Regional Research Ethics Committee Region Midtjylland)
Record Dates: First submitted 2024-01-02; First posted 2024-01-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples stored for batch analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ALS patients: Patients enrolled prior to determination of diagnosis on referral to neurophysiological examination. When the diagnosis is later established they get categorized as ALS patients.
  ALS patients with recent diagnosis might also be included directly.
  Interventions: Other: Observational study
- ALS mimic disease patients: Patients enrolled prior to determination of diagnosis on referral to neurophysiological examination. When diagnosis is later established and the diagnosis is NOT ALS they get categorized as ALS mimic disease patients.
  Interventions: Other: Observational study
- Healthy controls: Healthy controls.
  Interventions: Other: Observational study
- Disease controls: Patients with another motor neuron disease than ALS with slow progression.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Observational study.

SUMMARY:
The aim of this study is to describe the changes in the neuromuscular connection in patients with amyotrophic lateral sclerosis (ALS). The study consist of three substudies that have the following main hypothesis:

1. that ALS patients do not demonstrate equal capacity for muscle reinnervation and that reinnervation preserves muscle function and thereby slows down progression.
2. that blood concentrations of c-terminal agrin fragment (bCAF) reflect neuromuscular transmission deficiency and that blood concentration of neural cell adhesion molecule reflects degree of muscle denervation in patients.
3. that ALS patients with decrement when examined with repetitive nerve stimulation have more physical fatigue, slower progression, higher degree of reinnervation and higher bCAF compared to ALS patients without decrement.

There will be 3 inclusion groups.

1. patients referred for neurophysiological examination on suspicion of motor neuron disease.
2. healthy controls
3. disease control: patients with another motor neuron disease with slow progression.

All participants will be invited for at least 1 visit (baseline). If participants in group 1 eventually receive the diagnosis of ALS they will be invited for 2 additional visits 4 og 8 months after baseline visit, respectively.

Examinations will consist of:

* nerve conduction study
* repetitive nerve stimulation (except for healthy controls) to examine impairment of the neuromuscular connection.
* motor unit number estimation with MScanFit to estimate number and size of motor units.
* ultrasound examination of muscles to measure size and condition of muscles.
* questionnaires on fatigue and functional status.
* blood sample for measurement of specialized analysis (c-terminal agrin fragment and neural cell adhesion molecule) and routine analysis (liver and kidney function as well as neurofilament light chain)
* muscle strength assessment manually and by dynamometer to follow progression of muscle weakness
* bioelectrical impedance measurement to follow the overall body composition.

ELIGIBILITY:
Inclusion Criteria:

* Referred to clinical neurophysiological examination on suspicion of motor neuron disease or diagnosed with ALS according to Gold Coast criteria within the last 3 months.
* Age ≥18 years old
* Able and willing to provide informed consent

Exclusion Criteria:

* Former central or peripheral nervous system disease
* Diabetes
* Electrophysiological signs of polyneuropathy at baseline visit
* Pacemaker
* Pregnancy

For disease controls the exclusion criteria are the same, but the inclusion criteria:

* Diagnosed with disease with slow, progressive loss of motor neurons
* Age ≥18 years old
* Able and willing to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients refered for neurophysiological examination or patients followed at out-patient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reinnervation | From baseline and 8 months
  Difference between fast and slow progressing patients in change in mean amplitude size of motor units as estimated by MScanFit motor unit number estimation.
Blood biomarkers | Baseline
  Difference in blood concentration of c-terminal agrin fragment and neural cell adhesion molecule at baseline between ALS patients, healthy controls and ALS mimic disease patients.
Fatigue and decrement | Baseline
  Difference in proportion of participants with decrement between ALS patients and ALS mimic disease patients as well as degree of fatigue among ALS patients with and without neuromuscular transmission deficiency.

OTHER OUTCOMES:
Difference in mean amplitude size over time in patients. | Baseline, 4 months and 8 months.
  Mean amplitude size measured by MScanFit technique.
Difference in motor unit number estimation over time in patients. | Baseline, 4 months and 8 months.
  Motor unit number estimation measured by MScanFit technique.
Difference in mean amplitude size between patients and control groups | Baseline.
  Mean amplitude size measured by MScanFit technique.
Muscle strength assessed with manual muscle strength testing | Baseline, 4 months and 8 months.
  Difference in measures from manual muscle strength testing.
Difference in isometric ankle dorsiflexion strength measured on dynamometer. | Baseline, 4 months and 8 months.
  Measured on dynamometer.
Difference in handgrip strength measured on dynamometer. | Baseline, 4 months and 8 months.
  Measured with handgrip dynamometer.
Correlation between decrement at repetitive nerve stimulation and signs of reinnervation as measured by mean amplitude size. | Baseline, 4 months and 8 months.
  Decrement measured with repetitive nerve stimulation and mean amplitude size measured with MScanFit technique.
Blood concentration of c-terminal agrin fragment and neural cell adhesion molecule. | Baseline, 4 months and 8 months.
  Difference in blood measurements of c-terminal agrin fragment, neural cell adhesion molecule, neurofilament light chain and routine kidney and liver markers.
Difference in muscle thickness as measured by ultrasound examination of muscles | Baseline, 4 months and 8 months.
  Measured by ultrasound examination.
Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised scores | Baseline, 4 months and 8 months.
  Difference in scores from Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised. Scale 0-48, with 48 being the best.
Multidimensional Fatigue Inventory scores | Baseline, 4 months and 8 months.
  Difference in scores from Multidimensional Fatigue Inventory. Scale 4-20, with 20 indicating worst degree of fatigue.
Fatigue Severity Scale scores | Baseline, 4 months and 8 months.
  Difference in scores from Fatigue Severity Scale. Scale 9-63, with 63 indicating worst degree of fatigue.
Difference in free fatt mass as measured by bioelectrical impedance analysis. | Baseline, 4 months and 8 months.
  Measured by bioelectrical impedance analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper H Storgaard, MD, Principal Investigator — Aarhus University and Department of Neurology, Aarhus University Hospital
Locations (1):
- Department of Neurology, Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No